CLINICAL TRIAL: NCT02420015
Title: Mobile Health Technology to Enhance Abstinence in Smokers With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00061683
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia; Cigarette Smoking
MeSH Terms: conditions — Schizophrenia; Cigarette Smoking | interventions — Nicotine Replacement Therapy; Nicotine Chewing Gum; Transdermal Patch; Nebulizers and Vaporizers; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- iCOMMIT (Experimental): The components of the intervention include 1) behavioral therapy in the form of mobile contingency management (mCM) designed to increase early abstinent rates; 2) pharmacotherapy for smoking cessation [including nicotine replacement therapy (NRT) and bupropion]; 3) four sessions of guideline based cognitive-behavioral smoking cessation counseling designed to increased coping skills specific to smoking cessation; 4) a smart-phone based relapse prevention application (the Stay Quit Coach) that is populated during the counseling sessions; and 5) SMS text messaging reminders to increase medication adherence.
  Interventions: Drug: Nicotine replacement therapy; Drug: Bupropion; Behavioral: cognitive-behavioral smoking cessation counseling; Behavioral: Mobile Contingency Management; Behavioral: Stay Quit Coach; Behavioral: SMS text messaging
- Control Group (Active Comparator): The components of the intervention include 1) pharmacotherapy for smoking cessation [including nicotine replacement therapy (NRT) and bupropion]; and 2) four sessions of guideline based cognitive-behavioral smoking cessation counseling designed to increased coping skills specific to smoking cessation.
  Interventions: Drug: Nicotine replacement therapy; Drug: Bupropion; Behavioral: cognitive-behavioral smoking cessation counseling

INTERVENTIONS:
Drug: Nicotine replacement therapy — Participants will be prescribed NRT patch and one nicotine rescue method (e.g., nicotine gum, lozenge, inhaler) for use during the post-quit phase of the study. Participants will be given the choice between nicotine gum, nicotine inhaler, or nicotine nasal spray, and will be instructed to use the rescue method as needed to reduce cigarette cravings
  Other Names: nicotine gum, patch, inhaler, and/or lozenge
Drug: Bupropion — All participants who are medically eligible will be prescribed bupropion, which they will start two weeks prior to their quit day. Dosage will be 150 mg/daily for days 1-7 and 300 mg/daily (administered in two daily doses) until the 3-month follow-up
  Other Names: Zyban
Behavioral: cognitive-behavioral smoking cessation counseling — Participants will receive four 20-minute smoking cessation counseling sessions and a participant manual. The four sessions are based on standard cognitive-behavioral therapy techniques shown to be efficacious for smoking cessation.
Behavioral: Mobile Contingency Management — Participants will be asked to provide video recordings of themselves taking carbon monoxide readings in order to confirm smoking abstinence. Participants are asked to upload these videos to the study's secured server, and are provided monetary reward for videos that suggest smoking abstinence.
  Other Names: mCM
  Arms: iCOMMIT
Behavioral: Stay Quit Coach — Stay Quit Coach is a smart phone application that serves as a source of readily available support and information for adults who are already in treatment to quit smoking and to help them stay quit after treatment. The app guides user in creating tailored plans that include their personal reasons for quitting, interactive tools to help users cope with urges to smoke, motivational messages, support contacts to help users stay smoke free and how to address lapses. Participants assigned to this condition will be asked to use Stay Quit Coach from Session 2 through the 6-month follow-up.
  Arms: iCOMMIT
Behavioral: SMS text messaging — Patients assigned to this condition will receive text messages relevant to their current status in their smoking quit attempt, including messages reminding participants to take their smoking cessation medication.
  Other Names: texting
  Arms: iCOMMIT

SUMMARY:
This study is designed to evaluate if a treatment the investigators call iCOMMIT is effective at helping smokers with schizophrenia stop smoking. iCOMMIT is a smoking cessation treatment that combines mobile technology with behavioral strategies, counseling, and medications.

DETAILED DESCRIPTION:
The purpose of this 2-arm randomized controlled trial (RCT) is to evaluate the efficacy of Multi-Component Mobile-enhanced Treatment for Smoking Cessation (iCOMMIT) in helping individuals with schizophrenia or other psychotic disorders stop smoking. Eligible participants will be randomized to receive iCOMMIT, which includes smoking cessation counseling, pharmacotherapy, and mobile technology components, or a control intervention that includes smoking cessation counseling and pharmacotherapy, but no mobile technology components. The control condition represents an intensive standard of care and helps control for monitoring, counselor, time, and attention effects.

The primary outcome for the study will be self-reported and bio-verified prolonged smoking abstinence at the 6-month follow-up. Self-reported prolonged abstinence will be verified by saliva cotinine assay. Secondary outcomes will include 7- and 30-day point prevalence abstinence at each assessment, where abstinence is defined as no tobacco use in the prior 7 or 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Currently smoke at least ten cigarettes a day
* Have been smoking for at least one year
* Meet criteria for schizophrenia, schizoaffective disorder, or another psychotic disorder based on structured clinical interview
* Can speak and write fluent conversational English
* Are between 18 and 70 years of age
* Are willing to make a smoking cessation attempt
* Score 26 or higher on the Montreal Cognitive Assessment

Exclusion Criteria:

* Have a history of myocardial infarction in the past 6 months
* Have a contraindication to NRT with no medical clearance from the primary care provider or study physician
* Use and unwillingness to stop use of other forms of nicotine such as cigars, pipes, or chewing tobacco
* Are pregnant
* Meet criteria for a current manic episode based on structured clinical interview
* Are currently enrolled in another smoking cessation trial
* Are currently imprisoned or in psychiatric hospitalization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean C Beckham, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was deemed ineligible to participate in the study prior to randomization because that participant couldn't read or write English.
Groups:
- iCOMMIT: Components include:
  1. mobile contingency management (mCM): Participants provide video recordings of themselves taking carbon monoxide readings to confirm smoking abstinence.
  2. pharmacotherapy for smoking cessation: Includes nicotine replacement therapy [nicotine patch and one nicotine rescue method (e.g., nicotine gum, lozenge, inhaler)] and bupropion (150 mg/daily for days 1-7 and 300 mg/daily thereafter)
  3. 4 sessions cognitive-behavioral smoking cessation counseling;
  4. Stay Quit Coach: Stay Quit Coach is a smart phone application that provides support and information for adults who are already in treatment to quit smoking and to help them stay quit after treatment.
  5. SMS text messaging: Patients assigned to this condition will receive text messages relevant to their current status in their smoking quit attempt.
- Control Group: Components include:
  1. pharmacotherapy for smoking cessation: Includes nicotine replacement therapy [nicotine patch and one nicotine rescue method (e.g., nicotine gum, lozenge, inhaler)] and bupropion (150 mg/daily for days 1-7 and 300 mg/daily thereafter)
  2. 4 sessions cognitive-behavioral smoking cessation counseling;
Period: Overall Study
Arm/Group | iCOMMIT | Control Group
Started | 21 | 13
Completed | 21 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iCOMMIT | Control Group | Total
Number analyzed (Participants) | 21 | 13 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.24 (10.30) | 46.92 (10.30) | 48.39 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 13 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 6 | 19
  White | 3 | 1 | 4
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 21 | 13 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Self-report Prolonged Abstinence
Description: Prolonged abstinence will exclude tobacco use in the first two weeks following the quit date, as is consistent with other smoking cessation trials.
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | iCOMMIT | Control Group
Number analyzed (Participants) | 21 | 13
Participants | 6 | 3

2. Primary Outcome: Number of Participants Whose Prolonged Abstinence is Bio-verified
Description: Self-reported prolonged abstinence (primary outcome) will be verified by cotinine assay. Saliva samples will be collected from participants who self-report prolonged abstinence at each follow-up.
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | iCOMMIT | Control Group
Number analyzed (Participants) | 21 | 13
Participants | 3 | 2

3. Secondary Outcome: Number of Participants Who Report 7 Day Point Prevalence Abstinence
Description: Secondary smoking outcomes will include 7-day point prevalence abstinence at each assessment, where abstinence is defined as no tobacco use in the prior 7 days.
Time Frame: 3 months post-quit attempt (Session 5)
Measure: Count of Participants; unit: Participants
Arm/Group | iCOMMIT | Control Group
Number analyzed (Participants) | 21 | 13
Participants | 2 | 1

4. Secondary Outcome: Number of Participants Who Report 30 Day Point Prevalence Abstinence
Description: Secondary smoking outcomes will include 30-day point prevalence abstinence at each assessment, where abstinence is defined as no tobacco use in the prior 30 days.
Time Frame: 3 months post-quit attempt (Session 5)
Measure: Count of Participants; unit: Participants
Arm/Group | iCOMMIT | Control Group
Number analyzed (Participants) | 21 | 13
Participants | 2 | 1

5. Secondary Outcome: Number of Participants Who Report 7 Day Point Prevalence Abstinence
Description: as for outcome 3
Time Frame: 6 months post-quit attempt (Session 6)
Measure: Count of Participants; unit: Participants
Arm/Group | iCOMMIT | Control Group
Number analyzed (Participants) | 21 | 13
Participants | 4 | 2

6. Secondary Outcome: Number of Participants Who Report 30 Day Point Prevalence Abstinence
Description: as for outcome 4
Time Frame: 6 months post-quit attempt (Session 6)
Measure: Count of Participants; unit: Participants
Arm/Group | iCOMMIT | Control Group
Number analyzed (Participants) | 21 | 13
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Data were collected for approximately nine months (from the baseline visit to the 6-month follow-up visit).
Arm/Group | iCOMMIT | Control Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/21 | 3/13
Other Adverse Events (participants affected / at risk) | 13/21 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iCOMMIT (N=21) | Control Group (N=13)
Hospitalization (Psychiatric disorders) | 2 (2) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iCOMMIT (N=21) | Control Group (N=13)
Suicidal ideation (Psychiatric disorders) | 3 (4) | 1 (1)
Mouth and/or throat irritation (General disorders) | 3 (3) | 2 (2) — study-related
Altercation with police (Social circumstances) | 0 (0) | 1 (1)
Jitteriness, shakiness (Nervous system disorders) | 2 (2) | 1 (1) — Related to bupropion use
Sleep problems and/or nightmares (Psychiatric disorders) | 3 (4) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Related to nicotine patch use
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Related to quitting smoking
Family violence (Social circumstances) | 2 (2) | 0 (0) — Not related to study participation
Rape (Social circumstances) | 0 (0) | 1 (1) — Not related to study participation
Increased psychiatric symptoms (Psychiatric disorders) | 1 (2) | 1 (1) — Not related to study procedures, includes increased hallucinations and/or depressed mood
Nausea, upset stomach (Gastrointestinal disorders) | 2 (2) | 5 (5)
Flu (General disorders) | 2 (2) | 1 (1) — Not study related
dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Car accident (Social circumstances) | 1 (1) | 0 (0)
Death in family (Social circumstances) | 0 (0) | 1 (1)
Eye infection (Eye disorders) | 0 (0) | 1 (1)
Increased foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Related to pre-existing medical conditions
Benign tumor removed from lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pre-existing medical condition
Dental surgery (Surgical and medical procedures) | 1 (2) | 0 (0) — Related to pre-existing medical condition
Pain (General disorders) | 1 (1) | 0 (0) — Related to pre-existing medical condition
Increased seizures (Nervous system disorders) | 1 (2) | 0 (0) — Related to pre-existing medical condition
Swelling in leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Related to pre-existing medical condition

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT02420015/Prot_SAP_000.pdf